CLINICAL TRIAL: NCT05493956
Title: A Randomised Study of Consolidation CTRT Versus Observation After First Line Chemotherapy in Advanced Gallbladder Cancer: RACE-GB Study
Brief Title: A Randomised Study of Consolidation CTRT Versus Observation After First Line Chemotherapy in Advanced Gallbladder Cancer
Acronym: RACE-GB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-30-IP-108
Record Dates: First submitted 2022-08-03; First posted 2022-08-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Gallbladder Cancer Unresectable
MeSH Terms: interventions — Chemoradiotherapy; Observation

STUDY DESIGN:
Intervention Model Description: Consolidation chemoradiation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consolidation chemoradiation (Experimental): 6 cycles of Chemotherapy with Gemcitabine and Cisplatin will be followed by Concurrent Chemo-radiation with capecitabine
  Interventions: Radiation: chemoradiation
- Observation (Active Comparator): 6 cycles of Chemotherapy with Gemcitabine and Cisplatin will be followed by observation
  Interventions: Radiation: chemoradiation

INTERVENTIONS:
Radiation: chemoradiation — Radiation dose of 54 Gy will be given alongwith concurrent capecitabine
  Other Names: Observation

SUMMARY:
This will be a phase III randomized trial of advanced gall bladder cancers. 140 patients will be randomized. Randomisation will be on a 1:1 ratio between the experimental arm and the control arm.

Observation Arm : 6 cycles of Chemotherapy with Gemcitabine and Cisplatin will be followed by observation Chemotherapy followed by Chemo-radiotherapy Arm (CTRT): 6 cycles of Chemotherapy with Gemcitabine and Cisplatin will be followed by Concurrent Chemo-radiation with capecitabine (experimental arm).

DETAILED DESCRIPTION:
Treatment:

Chemotherapy followed by Chemo-radiotherapy:

Patients in experimental arm will be administered 6 cycles of gemcitabine 1000 mg/m2 d 1+8 and cisplatin 25mg/m2 d 1+8 repeated 3 weekly followed by abdominal radiotherapy using a standardized 3 dimensional conformal radiotherapy (3DCRT) technique on a linear accelerator operating at beam energy of >= 6MV.The total target dose of RT will be 45Gy in 25 fractions of 1.8 Gy to GBC and lymphatics (GBC, liver infiltration, periportal coeliac, superior mesenteric and paraortic lymphnodes till L2) followed by a boost of 9 Gy to the GBC. GBC mass alongwith liver infiltration would be GTV, and a 5mm margin around it would be GB_CTV. Nodal CTV would be delineated after combining PV, CA, SMA and aortic nodes. A Boolean of GB_CTV and Nodal CTV would be Final CTV. PTV margin would be 1 cm around Final CTV. DVH constraints would be : mean liver dose<30 Gy (liver would be delineated after subtracting GB_CTV), mean kidney dose <18 Gy (combining both kidneys). Other OAR to be delineated: stomach, bowel and their doses to be noted. Concurrent capecitabine to be given @1250 mg/m2 (Monday to Friday). Weekly clinical ,haemogram, LFT assessments will be done during the treatment.

Toxicities documented during adjuvant therapy will be recorded using the CTCAE version 3.0 (NCI 2006 scale). Toxicities arising more than 90 days since the completion of radiation therapy and attributed to radiation will be assessed according to CTCAE criteria and counted as late radiation toxicities.

Observation : enrolled patients will be administered 6 cycles of gemcitabine 1000 mg/m2 d 1+8 and cisplatin 25mg/m2 d 1+8 repeated 3 weekly for 6 cycles and then kept on observation.

QOL forms would be taken at baseline (before randomization, 2nd week RT and one week after completion of RT.)

Follow-up:

Interim analysis will be done at 50% recruitment or at 1.5 years of study whichever is earlier. After completion of treatment patients will be followed up and assessed clinically every month till disease progression. A CECT abdomen at 2 months would be done to assess response to treatment. Patients who develop symptoms of disease progression would be advised CECT scan to confirm disease progression before administering second-line chemotherapy (CAPIRI). Quality of Life assessment: This will be done using FACT hepatic scale at the time of randomization, second week of radiotherapy and one month after completion of radiotherapy.

In the control arm it will be assessed at the time of randomization, and at one month and 3 months of follow-up. Sample size estimation Assuming 2 year survival probability of the patients were 0.25 and 0.08 in the treatment (group1) and control (group2), at minimum two sided 95% confidence interval and 80% power of the study, overall sample size came out to be 132 subjects (66 in the group1 and 66 in the group2) using a two-sided log rank test. The proportion dropping out in each of the treatment and control group was 0.10 (ie10%). The proportion of switching from the treatment to control or control to treatment is assumed to be Nil.

Therefore in this study 70-70 patients will be included in the treatment and control groups (total 140).

Sample size was estimated using power analysis and sample size version-8 (PASS-2008).

ELIGIBILITY:
Inclusion Criteria:

* Rt hepatic artery involvement
* Rt Branch of portal vein and main PV involvement
* CBD/CHD/primary biliary confluence involvement
* Duodenum, pancreas, colon involvement
* omental metastases, liver involvement limited to segment 4,5
* Nodes in the hepato-duodenal, peripancreatic, common hepatic artery region, Para or preaortic region
* Good performance status
* BMI >15
* Have normal organ and marrow function

Exclusion Criteria:

* Multiple liver Metastasis as evident on CT scan abdomen .
* Presence of ascites
* Presence of jaundice (obstructive jaundice)
* Poor performance status (KPS<70)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | one year
  Time from diagnosis to death

SECONDARY OUTCOMES:
Progression free survival | one year
  time from diagnosis to evidence of disease progression
Toxicity due to consolidation chemoradiation | 24 weeks
  Toxicity during and after completion of chemo-radiotherapy
Hepatobiliary symptom index | 24 weeks
  Hepatobiliary symptom index ((physical, social, emotional and functional well being according to Fact-hep score)

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Agrawal, MD, Principal Investigator — SGPGIMS
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No